CLINICAL TRIAL: NCT06892249
Title: Suitability of Two Flavours of a High-energy, Low-protein Formula (Renalive® LP) in Chronic Kidney Disease Stage 3b-5 Outpatients in Taiwan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi Taiwan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rena-001-CEN
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: CKD; Low Protein Dietary Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Renalive® LP (Experimental)
  Interventions: Dietary Supplement: Renalive® LP, flavour Vanilla; Dietary Supplement: Renalive® LP, flavour Cappuccino

INTERVENTIONS:
Dietary Supplement: Renalive® LP, flavour Vanilla — flavour Vanilla
Dietary Supplement: Renalive® LP, flavour Cappuccino — flavour Cappuccino

SUMMARY:
Purpose of study To evaluate suitability of two flavours of a high energy low protein formula (Renalive® LP) as oral nutritional supplement and meal replacement in chronic kidney disease stage 3b-5 outpatients Inclusion criteria (1) Diagnosed with chronic kidney disease stage 3b-5 (with history of eGFR<45 mL/min/1.73 m2) (2) Age: 18-80 years (3) Outpatients with instruction to keep a low protein diet (0.55-0.8 g protein /kg actual body weight/ day) in the last 3 months as evaluated by the Investigator.

(4) Written Informed Consent from patient. Exclusion criteria

1. Has received dialysis or are expected to start dialysis within the next 3 months.
2. Patients awaiting kidney transplant.
3. Body mass index (BMI) <18 kg/m2 or BMI >30 kg/m2
4. Malnourished patients with albumin <3 g/dL in need of extra calories and nutrients
5. Patients receiving or having received oral/enteral/parenteral nutrition supplementation for special medical purpose in the last 28 days
6. Severe liver disease, malignant neoplastic disease, current significant infectious disease (apart from flu, cold, Hepatitis C virus (HCV) carrier, Hepatitis B virus (HBV) carrier, skin infection) deemed unsuitable for entering the trial as evaluated by the Investigator
7. Existing gastrointestinal disease or pathological findings that cannot tolerate enteral nutrition or render enteral nutrition unfeasible, such as shock, acute upper gastrointestinal bleeding, intestinal sluggishness, intestinal obstruction, or malabsorption, such as inflammatory bowel disease, pancreatic disease, or gastrointestinal surgery
8. Severe impairment of gastrointestinal function, i.e. severe constipation or acute diarrhoea (≥3 loose or watery stools a day)
9. Swallowing difficulty or high risk of aspiration
10. Central nervous system and/or certain psychiatric disorders where the patient is considered as not yet clinically stable and/or not suitable to participate in this study by the Investigator
11. Known allergic reaction or intolerance to any ingredient of the intervention formula.
12. Surgery or hospitalization scheduled during the trial
13. Suspected drug abuse
14. Unable to follow study instructions or keep a dietary diary
15. Pregnant or lactating women
16. Participation in other clinical trials using investigational drugs within 30 days before the start of the trial or during the trial.

Primary Endpoint

(1) Change in body weight from Baseline to end of treatment at Week 4 (Week 4 - Baseline) Secondary Endpoints

1. Daily dietary intake of energy, protein, sodium, potassium, magnesium, phosphorus, and calcium at Baseline, Week 2 and 4 based on a 3-Day Dietary Record
2. Change of nutritional status using body weight, BMI, and body composition as indicators:

   * Change in body weight from Baseline to Week 2
   * Change in BMI from Baseline to Week 2 and week 4
   * Change in body composition from Baseline to Week 4 using bioelectrical impedance assessment
3. Change of the physical performance using hand grip strength as an indicator from Baseline to Week 4
4. Change of renal function:

   * Change in estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) from Baseline to Week 4
   * Change in blood urea nitrogen and serum creatinine from Baseline to Week 2 and 4
5. Serum albumin and pre-albumin at Baseline and Week 4
6. Blood electrolytes (sodium, potassium, phosphorus, calcium, magnesium) at Baseline, Week 2 and 4
7. Serum C-reactive protein (CRP) at Baseline, Week 2 and 4
8. Compliance rate (%) to Renalive® LP

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with chronic kidney disease stage 3b-5 (with history of eGFR<45 mL/min/1.73 m2)
2. Age: 18-80 years
3. Outpatients with instruction to keep a low protein diet (0.55-0.8 g protein /kg actual body weight/ day) in the last 3 months as evaluated by the Investigator
4. Written Informed Consent from patient

Exclusion Criteria:

1. Has received dialysis or are expected to start dialysis within the next 3 months
2. Patients awaiting kidney transplant
3. Body mass index (BMI) <18 kg/m2 or BMI >30 kg/m2
4. Malnourished patients with albumin <3 g/dL in need of extra calories and nutrients
5. Patients receiving or having received oral/enteral/parenteral nutrition supplementation for special medical purpose in the last 28 days
6. Severe liver disease, malignant neoplastic disease, current significant infectious disease (apart from flu, cold, Hepatitis C virus (HCV) carrier, Hepatitis B virus (HBV) carrier, skin infection) deemed unsuitable for entering the trial as evaluated by the Investigator
7. Existing gastrointestinal disease or pathological findings that cannot tolerate enteral nutrition or render enteral nutrition unfeasible, such as shock, acute upper gastrointestinal bleeding, intestinal sluggishness, intestinal obstruction, or malabsorption, such as inflammatory bowel disease, pancreatic disease, or gastrointestinal surgery
8. Severe impairment of gastrointestinal function, i.e. severe constipation or acute diarrhoea (≥3 loose or watery stools a day)
9. Swallowing difficulty or high risk of aspiration
10. Central nervous system and/or certain psychiatric disorders where the patient is considered as not yet clinically stable and/or not suitable to articipate in this study by the Investigator
11. Known allergic reaction or intolerance to any ingredient of the intervention formula
12. Surgery or hospitalization scheduled during the trial
13. Suspected drug abuse
14. Unable to follow study instructions or keep a dietary diary
15. Pregnant or lactating women
16. Participation in other clinical trials using investigational drugs within 30 days before the start of the trial or during the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from Baseline to end of treatment at Week 4 (Week 4 - Baseline) | 4 weeks

SECONDARY OUTCOMES:
Daily dietary intake of energy, protein, sodium, potassium, magnesium, phosphorus, and calcium at Baseline, Week 2 and 4 based on a 3-Day Dietary Record | 4 weeks
Change in BMI from Baseline to Week 2 and Week 4 | 4 weeks
Change in body composition from Baseline to Week 4 using bioelectrical impedance assessment | 4 weeks
Change of the physical performance using hand grip strength as an indicator from Baseline to Week 4 | 4 weeks
Change in estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) from Baseline to Week 4 | 4 weeks
Change in blood urea nitrogen and serum creatinine from Baseline to Week 2 and 4 | 4 weeks
Serum albumin and pre-albumin at Baseline and Week 4 | 4 weeks
Blood electrolytes (sodium, potassium, phosphorus, calcium, magnesium) at Baseline, Week 2 and 4 | 4 weeks
Serum C-reactive protein (CRP) at Baseline, Week 2 and 4 | 4 weeks
Compliance rate (%) to Renalive® LP | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan, Taiwan